CLINICAL TRIAL: NCT00906477
Title: Intensive Training of Arm and Hand Function in People With Stroke - A Randomized Controlled Multisite Trial.
Brief Title: Norwegian Constraint-Induced (CI) Therapy Multisite Trial
Acronym: NORCIMT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was extended for 2.5 years. A further extension could not be funded. When the study was halted in June 2012, 47 subjects were included.
Sponsor: University Hospital of North Norway (Other)
Collaborators: Helse Nord (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Helse Nord SAT 544-06
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early intervention (Experimental): Modified CI therapy starting between 7 and 28 days post stroke.
  Interventions: Procedure: Modified CI therapy
- Delayed intervention (Active Comparator): Modified CI Therapy starting 6 months post stroke
  Interventions: Procedure: Modified CI therapy

INTERVENTIONS:
Procedure: Modified CI therapy — 10 treatment days 3 hours a day: Shaping exercises 2 hours. Task practice 0,5 hours. Behavioral therapy (Transfer package) 0,5 hour. Encouragement to wear a restraining mitt on the least affected arm for all safe activities.
  Other Names: Constraint induced movement therapy; Modified constraint induced movement therapy; CIMT; mCIMT; Forced use therapy

SUMMARY:
The purpose of this study is to determine whether modified CI therapy treatment is suitable and effective in the early rehabilitation after stroke, and to compare early CI intervention with a later CI intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Stroke at more than 5 and less than 26 days ago.(Either first stroke or second stroke without detectable arm weakness after the first stroke).
* Modified ranking scale 0-2 before admission
* Persistent unilateral arm or hand paresis (Scandinavian Strokes scale (SSS) arm motor function 2-5 or SSS hand motor function 2-4)
* Able to lift two fingers with the forearm pronated on the table or able to extend the wrist at least 10 degrees from fully flexed position.
* Able to follow a two step command.
* Mini Mental State examination score of more than 20 (or more than 16 in combination with expressive aphasia)

Exclusion Criteria:

* Modified Rankin Scale > 4
* Unable to give informed consent
* Large hemispatial neglect (more than two cm on the Line Bisection Test)
* Not expected to survive one year due to other illnesses (eg cardiac, malignancy)
* Injury or condition in the affected upper extremity that limited use prior to the stroke.
* Other neurological condition affecting motor function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-10; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Wolf Motor function test | 6 months post inclusion

SECONDARY OUTCOMES:
Arm use accelerometry | 6 months
Fugl Meyer Motor Assessment | 6 months
Nine hole peg test | 6 months
Wolf Motor Function Test | 12 months
Arm use accelerometry | 12 months
Fugl Meyer Motor Assessment | 12 months
Nine Hole Peg Test | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gyrd Thrane, Cand. San., Principal Investigator — University Hospital of North Norway; Audny GM Anke, MD, PhD, Study Chair — University Hospital of North Norway; Bent Indredavik, MD, PhD, Principal Investigator — Trondheim University Hospital; Torunn Askim, PhD, Principal Investigator — Norwegian University of Technology and Science; Roland Stock, MSc, Principal Investigator — Trondheim University Hospital
Locations (5):
- Norway (5):
  - Trondheim University Hospital, Trondheim, Sør-Trøndelag
  - University Hospital of North Norway, Tromsø, Troms
  - Levanger Hospital, Levanger
  - Oslo University hospital, Aker, Oslo
  - Vestfold Klinikk Fysikalske medisin og rehabilitering, Kysthospital, Stavern

REFERENCES:
- [Derived] Thrane G, Askim T, Stock R, Indredavik B, Gjone R, Erichsen A, Anke A. Efficacy of Constraint-Induced Movement Therapy in Early Stroke Rehabilitation: A Randomized Controlled Multisite Trial. Neurorehabil Neural Repair. 2015 Jul;29(6):517-25. doi: 10.1177/1545968314558599. Epub 2014 Nov 14. PMID 25398726